CLINICAL TRIAL: NCT06010511
Title: White Matter Hyperintensity Shape and Glymphatics
Acronym: WHIMAS
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Alzheimer Nederland (Unknown)
Responsible Party: Principal Investigator, Jeroen de Bresser, Principal Investigator; MD; PhD, Leiden University Medical Center
Other Study IDs: WHIMAS
Record Dates: First submitted 2023-07-18; First posted 2023-08-24 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Small Vessel Diseases; Dementia, Mixed; Dementia, Vascular; Mild Cognitive Impairment; Cognitive Impairment; Cognitive Decline
Keywords: dementia; cerebral small vessel disease; White matter hyperintensities; cognitive impairment; cognitive decline; Glymphatics
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Mixed Dementias; Dementia, Vascular; Cognitive Dysfunction; Dementia | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Memory clinic patients: We will prospectively include patients with memory complaints and/or vascular brain abnormalities (n=50; over 65 years of age) from the memory clinic (or geriatric clinic) at one of their first visits, prior to any diagnosis.
  Interventions: Other: 3T MRI scan; Other: 7T MRI scan; Behavioral: Neuropsychological assessment; Other: General baseline data

INTERVENTIONS:
Other: 3T MRI scan — Conventional (3T) brain MRI scans will be used to determine global and functional markers of cerebral SVD, like WMH volume and presence of lacunes, microbleeds and superficial siderosis (3D T1, 3D FLAIR, SWI, DWI), hemodynamics (arterial spin labelling & flow territory mapping) and white matter structural integrity (diffusion tensor imaging (DTI)). Furthermore, we want to measure structural integrity with a novel MR fingerprinting sequence and an inhomogeneous magnetization transfer (ihMT) MRI scan. We also want to apply a fMRI scan technique to measure CSF fluctuations in the 4th ventricle as a measure of brain glymphatics. Also the flow-territory mapping sequence is a non-standard sequence. Heart rate and respiratory signal will be measured during the scans (3T and 7T MRI) with standard vendor-supplied equipment.
Other: 7T MRI scan — Ultra-high field (7T) brain MRI scans will be used to determine WMH shape and other markers of cerebral SVD in or surrounding the WMH, like local enlarged perivascular spaces, (cortical) microinfarcts and microbleeds (T1, T2, FLAIR and T2*) and vascular pulsatility (phase contrast MRI). Moreover, a recently implemented MRI technique to measure glymphatic flow in perivascular spaces will be used.
Behavioral: Neuropsychological assessment — * Mini-mental state examination
  * Clock drawing
  * 15-Word Verbal Learning Test, immediate and delayed
  * Visual Association Test
  * Stroop Color Word Test, 40 item version
  * Trail Making Test A&B
  * Letter Digit Substitution Test
  * Animal fluency test
  * Hospital anxiety and depression scale
  * Informant Questionnaire on Cognitive Decline in the Elderly
Other: General baseline data — Baseline data, such as age, sex, psychiatric comorbidity and medication lists will be extracted from the patient files.
  Age (Year of birth); Years of education; BMI (height & weight); Sex; Verhage scale (education); Smoking status; Blood values; Sleep habits; Waste-hip ratio; Blood pressure; Current/general cardiovascular health; Psychiatric comorbidity; medical history related to cardiovascular health.

SUMMARY:
In a society with increased life expectancy, the economic, social and personal burden of dementia increases. Dementia is often caused by a combination of neurovascular and neurodegenerative diseases. Impaired brain clearance is suggested to be closely related to dementia development, as waste products (e.g. amyloid beta) accumulate in the brain, leading to neurodegeneration. Cerebral small vessel disease (SVD) is the most common neurovascular disease that even contributes to about 45% of dementia pathophysiology in patients with a diagnosis of Alzheimer's dementia. White matter hyperintensities of presumed vascular origin (WMH) are the key brain MRI manifestation of cerebral SVD. There is evidence that the currently known and MRI-visible WMH are landmarks of an already progressed stage of the underlying pathology. The pathophysiology of WMH has been attributed to multiple underlying mechanisms, such as hypoperfusion, defective cerebrovascular reactivity and blood-brain barrier dysfunction. Furthermore, different anatomical locations and different types of WMH are related to different underlying pathological changes. Using ultra-high field 7T MR imaging techniques WMH lesions can be detected with a higher sensitivity and resolution than on 3T MRI. The hypothesis is that different pathological mechanisms of cerebral SVD lead to variations in WMH shape. Moreover, the brain clearance ('glymphatic') system of the brain appears to be tightly connected to dementia pathology. Thus, novel markers of glymphatic activity could aid to describe and understand the pathology.

DETAILED DESCRIPTION:
Aim:

The overall aim is to study how different pathological mechanisms in cerebral SVD influence WMH shape.

Primary objective:

To study the association of a more complex WMH shape with abnormalities in small vessel morphology.

Secondary objectives:

To study the association between WMH shape and cognition/other cerebral small vessel disease markers. To study the association of novel MRI markers of glymphatics with cerebral SVD markers and cognition.

Study design: Cross-sectional study that will be conducted at the Leiden University Medical Center (LUMC). Patients will be included from the LUMC or the Alrijne Hospital Leiden. The study contains 3T and 7T MRI scans, as well as neuropsychological assessments. The data will be analyzed by performing association analysis.

Study population: Patients of the memory/geriatric clinic that are over 65 years of age.

Main study parameter/endpoint: In order to postulate underlying mechanisms related to WMH shape variations the investigators will study the association between a more complex WMH shape and structural and functional markers of cerebral SVD (such as lacunes and microbleeds).

WMH shape is assessed as follows: Convexity, solidity, concavity index, and fractal dimension are calculated for periventricular/confluent WMH. A lower convexity and solidity, and higher concavity index and fractal dimension indicate a more irregular shape of periventricular/confluent WMH. For deep WMH, fractal dimension and eccentricity are determined. A higher eccentricity and fractal dimension indicate a more complex shape of deep WMH.

Other study parameters: The investigators want to investigate WMH shape parameters and the association with cognition (mini-mental state exam, clinical dementia rating and cognitive domain scores). Another endpoint is to investigate if different WMH phenotypes can be identified (by machine learning models). Moreover, the association between SVD markers/cognition and novel glymphatics markers (such as size of perivascular spaces, CSF mobility and 4th ventricle CSF flow dynamics) will be investigated.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The participants will not directly benefit from the results of the study. However, their contribution to the study will add important information about the pathophysiology of the cerebrovascular pathology that contributes to dementia. Therefore, it is not possible to study the research question in a different population group. The ultra-high field 7T MRI system is widely used in a research setting and since its first introduction in the 1990s no serious adverse events have been reported. Important temporary side-effects are vertigo, nausea and involuntary eye motion due to forces on ion currents in the semicircular loops. As all MRI scans are performed within a maximum of 60 minutes and without any contrast agents, the participant burden is seen as a non-substantial burden.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the memory or the geriatric clinic of the LUMC, the Alrijne Hospital Leiden or the Haga Hospital the Hague
* From 65 years of age
* Eligible for MRI
* Native-level Dutch speaker

Exclusion Criteria:

* Claustrophobia
* Contraindications for MRI such as metal implants and pacemaker
* Use of benzodiazepines
* Initiated treatment with antidepressants less than 6 weeks prior to inclusion
* Not being able to provide written informed consent (assessed by the treating physician)
* Individuals that have been declared mentally incapacitated
* Other severe neurological disease besides dementia related
* Cognitive impairment due to known other neurological disease
* Previous brain surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: We will prospectively include patients with memory complaints and/or vascular brain abnormalities (n=50; over 65 years of age) from the memory clinic at one of their first visits, prior to any diagnosis, at the Leiden University Medical Center, the Alrijne Hospital Leiden or the Haga Hospital the Hague. If not enough eligible patients are available from the memory clinic, we will include participants from the geriatric clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
WMH shape | at study visit during inclusion up to 3 years
  The investigators will use an in-house developed analysis pipeline to calculate WMH shape on 3T and 7T brain MRI scans. Associations between WMH shape and other SVD markers and cognition will be investigated with linear and logistic regression (at least corrected for age and sex).

SECONDARY OUTCOMES:
Brain clearance | at study visit during inclusion up to 3 years
  Measured on brain MRI as a marker of glymphatic activity.
Perivascular space volume | at study visit during inclusion up to 3 years
  This marker will be measured on brain MRI.
WMH subtypes | at study visit during inclusion up to 3 years
  Based on WMH parameters the investigators will study if subtypes of WMH can be identified.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen de Bresser, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bos D, Wolters FJ, Darweesh SKL, Vernooij MW, de Wolf F, Ikram MA, Hofman A. Cerebral small vessel disease and the risk of dementia: A systematic review and meta-analysis of population-based evidence. Alzheimers Dement. 2018 Nov;14(11):1482-1492. doi: 10.1016/j.jalz.2018.04.007. Epub 2018 May 21. PMID 29792871
- [Background] Ghaznawi R, Geerlings MI, Jaarsma-Coes M, Hendrikse J, de Bresser J; UCC-Smart Study Group. Association of White Matter Hyperintensity Markers on MRI and Long-term Risk of Mortality and Ischemic Stroke: The SMART-MR Study. Neurology. 2021 Apr 27;96(17):e2172-e2183. doi: 10.1212/WNL.0000000000011827. Epub 2021 Mar 16. PMID 33727406
- [Background] Ghaznawi R, Geerlings MI, Jaarsma-Coes MG, Zwartbol MH, Kuijf HJ, van der Graaf Y, Witkamp TD, Hendrikse J, de Bresser J. The association between lacunes and white matter hyperintensity features on MRI: The SMART-MR study. J Cereb Blood Flow Metab. 2019 Dec;39(12):2486-2496. doi: 10.1177/0271678X18800463. Epub 2018 Sep 11. PMID 30204039
- [Background] Keller JA, Sigurdsson S, Klaassen K, Hirschler L, van Buchem MA, Launer LJ, van Osch MJP, Gudnason V, de Bresser J. White matter hyperintensity shape is associated with long-term dementia risk. Alzheimers Dement. 2023 Dec;19(12):5632-5641. doi: 10.1002/alz.13345. Epub 2023 Jun 12. PMID 37303267
- [Derived] Kuhn-Keller JA, Eiling I, Hirschler L, Vaclavu L, Witjes-Ane MN, Wijngaarden M, Nagtegaal M, Ercan E, Rius Ottenheim N, van der Elst M, Sohl E, van Buchem MA, Mooijaart S, van Osch MJ, de Bresser J. The White Matter Hyperintensity Shape and Brain Clearance (WHIMAS) Study for Identification of Novel 7T Magnetic Resonance Imaging Markers of Cerebral Small Vessel Disease: Protocol for a Cross-Sectional Study. JMIR Res Protoc. 2025 Dec 4;14:e77681. doi: 10.2196/77681. PMID 41344663